CLINICAL TRIAL: NCT01385228
Title: Phase I Study of Docetaxel, Prednisone and Pazopanib in Men With Metastatic Castrate-Resistant Prostate Cancer (mCRPC) and Poor-Risk Factors
Brief Title: Pazopanib, Docetaxel, Prednisone Prostate
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Daniel George, MD (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Sponsor-Investigator, Daniel George, MD, Associate Professor of Medicine, Duke University
Organization: Duke University (Other)
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Pro00026577; PZP113296 (Other Grant/Funding Number: GSK); c09-039 (Other: Prostate Cancer Clinical Trials Consortium)
Record Dates: First submitted 2011-06-12; First posted 2011-06-30 (Estimated); Last update posted 2018-06-06 (Actual); Status verified 2018-06

CONDITIONS: Prostate Cancer
Keywords: prostate cancer; metastatic; pazopanib; docetaxel; metastatic prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms; Neoplasm Metastasis | interventions — pazopanib; Docetaxel; Prednisone; pegfilgrastim

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Dose Level "Xa" (Experimental): once daily pazopanib for Days 1-21 in combination with docetaxel given IV on Day 1 and prednisone daily. Pegfilgrastim (Neulasta) every 21 days on Day 2, 3 or 4 of each cycle.
  Interventions: Drug: Pazopanib; Drug: Docetaxel; Drug: Prednisone; Drug: Pegfilgrastim
- Dose Level "Xb" (Experimental): once daily oral administration of pazopanib for Days 3-19 in combination with docetaxel given intravenous administration on Day 1 and prednisone daily. Pegfilgrastim (Neulasta) every 21 days on Day 2, 3 or 4 of each cycle.
  Interventions: Drug: Docetaxel; Drug: Pazopanib; Drug: Prednisone; Drug: Pegfilgrastim

INTERVENTIONS:
Drug: Pazopanib — Dose Level "Xa" - daily administration of pazopanib on days 1 through 21 starting at 400mg with a maximum dose of 1000mg.
  Other Names: Pazopanib (GW786034)
  Arms: Dose Level "Xa"
Drug: Docetaxel — Docetaxel given IV on Day 1 starting dose 60mg/m2 increase to 75mg/m2
  Other Names: Taxotere
Drug: Pazopanib — Dose Level "Xb" - daily administration of pazopanib on days 3 through 19 starting at 400mg with a maximum dose of 1000mg.
  Other Names: Pazopanib (GW786034)
  Arms: Dose Level "Xb"
Drug: Prednisone — 5mg Prednisone given twice daily days 1-21.
Drug: Pegfilgrastim
  Other Names: Neulasta

SUMMARY:
The primary purpose is to define the safety and tolerability of docetaxel/prednisone in combination with pazopanib (DPP) in men with metastatic Castration Resistant Prostate Cancer (mCRPC).

DETAILED DESCRIPTION:
This Phase I study will consist of a dose escalation portion which includes a dose escalation phase of 10 dose levels: (1a) docetaxel 60 mg/m2, pazopanib 400 mg daily, prednisone 5 mg BID; (2a) docetaxel 75 mg/m2, pazopanib 400 mg daily, prednisone 5 mg BID; and (3a) docetaxel 75 mg/m2, pazopanib 600 mg daily, prednisone 5 mg BID; (4a) docetaxel 75mg/m2, pazopanib 800 mg daily, (5a) docetaxel 75mg/m2, pazopanib 1000mg daily, prednisone 5 mg; (1b) docetaxel 60 mg/m2, pazopanib 400 mg daily x 17 days, prednisone 5 mg BID; (2b) docetaxel 75 mg/m2, pazopanib 400 mg daily x 17 days, prednisone 5 mg BID; and (3b) docetaxel 75 mg/m2, pazopanib 600 mg daily x 17 days, prednisone 5 mg BID; (4b) docetaxel 75mg/m2, pazopanib 800 mg daily x 17 days, (5b) docetaxel 75mg/m2, pazopanib 1000mg daily x 17 days, prednisone 5 mg. If the investigators see > 1 dose limiting toxicity (DLT) at Dose level 3 then the investigators would investigate docetaxel 75 mg/m2, pazopanib 600 mg daily, prednisone 5 mg BID (Dose level 3a). If < 1 DLT are seen at Dose level 3 and Pharmacokinetic (PK) analysis is complete and acceptable, then the investigators will proceed to dose level 4) docetaxel 75 mg/m2, pazopanib 1000 mg daily, prednisone 5 mg BID.

The investigators will dose escalate in a classic 3+3 design. The maximum tolerated dose (MTD) will be defined as the highest dose level that does not result in 2 or more dose limiting toxicities (DLTs). A dose expansion at the MTD of 10-15 patients (up to a total of 36 patients) will be accrued in order to further describe the safety profile.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed carcinoma of the prostate. Histologic evidence may be confirmed through local or metastatic biopsy review. Non-adenocarcinomas are permitted.
* Radiographic evidence of metastatic disease; non-evaluable, bone only metastasis is permitted.
* Evidence of disease progression despite castrate levels of testosterone (<50 ng/dl).
* At the time of screening, at least 2 weeks since prior palliative radiation therapy and 4 weeks from major surgery, and resolution of all toxic effects of prior therapy to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE); version 4.0 Grade < 1.
* Age >18 years
* Adequate laboratory parameters
* Eastern Cooperative Oncology Group (ECOG) performance status between 0 and 2
* Life expectancy greater than 3 months
* Written, signed and dated Institutional Review Board (IRB) approved informed consent form.

Exclusion Criteria:

* History of or active central nervous system metastases
* The use of immunologic, biologic, or hormonal therapies within 2 weeks of study entry.
* Major surgery, open biopsy, traumatic injury within 4 weeks of the screening visit
* Subjects who have not recovered from prior biopsy, surgery, traumatic injury, and/or radiation therapy.
* Previous treatment with docetaxel, including in the neo-adjuvant or adjuvant setting
* Presence of non-healing wound or ulcer
* Grade 3 or greater hemorrhage within the past month.
* Uncontrolled hypertension
* American Heart Association Class 2-4 heart disease or any history of congestive heart failure with an ejection fraction <40%, recent cardiovascular event (within 12 months) including unstable angina, any exertional angina, myocardial infarction, exertional or rest claudication, or stroke/Cerebral Vascular Event/Transient Ischemic Attack. Patients with known moderate to severe documented carotid or peripheral vascular disease are excluded. Angioplasty or stenting of coronary or peripheral arteries are exclusionary if within the past 12 months.
* Anticoagulation with warfarin (therapeutic doses of warfarin for catheter patency are permitted up to 2 mg/day). Low molecular weight heparin is permitted.
* Diabetes mellitus with glycosylated hemoglobin A1c (HbgA1c) > 8% despite therapy
* Subjects with active autoimmune disorder(s) being treated with systemic immunosuppressive agents within 4 weeks prior to the screening visit.
* Active infection(s), active antimicrobial therapy or serious intercurrent illness.
* Does not agree to use medically acceptable contraceptive methods while on study and for 3 months after the last dose of pazopanib.
* Any other major medical or psychiatric illness that, in the investigator's judgment, will substantially increase the risk associated with the subject's participation in this study, including inability to absorb oral medications.
* Known hypersensitivity to any of the components in the docetaxel infusion or other medical reasons for not being able to receive adequate premedication (for example, antihistamine or anti-inflammatory agents).
* CalculatedQT (QTc) interval on baseline EKG > 500milliseconds
* History or presence of nephrotic syndrome

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2011-06; Primary Completion 2015-07 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Number and Percent of Participants with Adverse Events as a Measure of Safety and Tolerability | 15 months
  The primary objective for the phase I study is to assess the safety and tolerability of pazopanib, docetaxel, and prednisone given in combination in patients with metastatic castration resistant prostate cancer.

SECONDARY OUTCOMES:
Establish the maximum tolerated dose | 15 months
  Determine the dose levels of pazopanib and docetaxel that are the most tolerated.
Establish the optimal dosing schedule | 15 months
  Establish the optimal dosing schedule for the combination of docetaxel, prednisone and pazopanib

CONTACTS AND LOCATIONS:
Overall Officials: Daniel J George, MD, Principal Investigator — Duke Cancer Institute
Locations (2):
- United States (2):
  - The University of Chicago, Chicago, Illinois
  - Duke Cancer Institute, Durham, North Carolina